CLINICAL TRIAL: NCT07125092
Title: A Study to Evaluate the Clinical Benefit and Safety of Medical Compression Garments in the Management of Patients With Lipœdema
Brief Title: A Study to Evaluate the Clinical Benefit and Safety of Medical Compression Garments in the Management of Patients With Lipedema
Acronym: LIP'EX
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Thuasne (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EC46 LIP'EX
Record Dates: First submitted 2025-07-28; First posted 2025-08-15 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Lipoedema
Keywords: lipoedema; compression; pain; quality of life
MeSH Terms: conditions — Lipedema; Pain

STUDY DESIGN:
Intervention Model Description: This is a prospective, open-label, study conducted over a period of 10 weeks in a population of patients with lipedema
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Compression group (Experimental): Compression device group:
  All patients enrolled in the study will be instructed to wear the compression garment for 8 weeks, as long as possible during the day.
  In parallel, all patients will receive the same advice about routine care: physical exercises, nutrition aspect that are part of the centre's current practice.
  Interventions: Device: compression group

INTERVENTIONS:
Device: compression group — All patients enrolled in the study will be instructed to wear the compression garment for 8 weeks, as long as possible during the day. In parallel, all patients will receive the same advice about routine care: physical exercises, nutrition aspect that are part of the centre's current practice.
  3 study visits are planned: the inclusion visit (V0) includes patient information and consent signature, measurements for custom-made compression stockings. The initial visit (V1) includes devices collection and fitting, patient questionnaires, physician assessment (medical and lipedema history, BMI, WHtR, blood sample collection, pain description, lipedema associated symptoms, leg perimeter measurements, Moisture Meter, pressure under the garment). The follow-up visit (V2) after 8 weeks includes: patient questionnaires and physician assessment.
  After 8 weeks, another compression garment will be given to the patient with a new satisfaction e-questionnaire at 10 weeks of follow-up.

SUMMARY:
Lipedema (LI) is a chronic condition, painful disease characterized by a disproportionate increase in adipose tissue and pain in women's legs and sometimes arms. Its prevalence is largely unknown, but lipedema is estimated to affect 0.06% to 11% of the female population. Even though this pathology is increasingly studied and working groups are collaborating to harmonize criteria, a crucial underlying problem of lipedema is the variability in identifying lipedema. Lipedema patients often suffer from obesity, physical disability and psychological impairments, and the effects on quality of life are significant. Almost all women with lipedema are dissatisfied with the disproportionality of their body and the stigma associated with it. In addition to weight gain, pain is one of the major symptoms of this pathology, but also limb heaviness, weakness, or difficulties with walking. Patients also tend to develop easy bruising, although these symptoms are not always present. Treatment of lipedema is aimed at relieving pain, maintaining/improving mobility, reducing volume of the limbs, and improving quality of life. It is important to note that compression therapy is one of the cornerstones of this treatment because of its anti-inflammatory effect on adipose tissue

DETAILED DESCRIPTION:
Wearing compression stockings leads to a significant reduction in oxidative stress, a finding that also indicates improved microcirculation in the subcutaneous tissue. Wearing compression stockings may relieve pain and may improve the ability of patients to move. In this context, the hypothesis is that the treatment of lipedema patients with compression stockings contributes to the reduction of lipedema-associated symptoms such as pain and heaviness and thus contributes to a better quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Lipedema diagnosed at least in the legs according to the initial Wold criteria modified by Herbst.
* Average pain in the legs over the last week ≥ 4 points on a 10 points Numerical Rating Scale visual analogue scale.
* Patient who has given his informed consent freely and signed it prior to any intervention in the study.

Exclusion Criteria:

* Patient for whom compression is contraindicated, such as untreated infections, skin irritation or lesions.
* Lipedema type I: Hips/buttocks.
* Patients who underwent liposuction.
* Patient with a WHtR higher than 0,58.
* Patient with active cancer, chemotherapy treatment, chronic inflammatory disease, chronic anti-inflammatory therapy (ex: TNF alpha).
* Patient with surgery scheduled/planned during the study period.
* Patient with a known allergy to the components used in the devices.
* Pregnant woman or woman of childbearing age without contraception.
* Patient currently participating in another clinical investigation that could impact the study endpoints.
* Patient with psychiatric, psychological, or neurological disorders that are incompatible with the proper follow-up of the clinical investigation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
Evolution of pain: Numeric Rating Scale (NRS) | Weekly between baseline and 8 weeks of follow-up
  The evolution of perceived leg pain (mean and maximum) related to lipedema is measured by Numeric Rating Scale (NRS). 0 corresponds to no pain and 10 to the maximum pain.

SECONDARY OUTCOMES:
Evolution of pain threshold under pressure (algometer) | From baseline to 8 weeks of follow-up
  The pain threshold under pressure is measured by an algometer. It is a non-invasive and painless instrument that consists of a dial, a cylinder attached to the dial, and a rod inside the cylinder, which ends in a 1 cm2 rubber tip.
Quality of life (QoL): Patient's opinion on Global Impression of Change (PGI-C) | 8 weeks
  The patient's impression of overall change is measured by the Patient's opinion on Global Impression of Change questionnaire (PGI-C). The scale has 7 levels of response :
  "no change or condition has got worse" that is the worst outcome (= 1 point) "almost the same, hardly any change at all" (= 2 points); "a little better , but no noticeable change" (= 3 points); "somewhat better, but the change has not made any real difference" (= 4 points); "moderately better, and a slight but noticeable change" (= 5 points); "better, and a definite improvement that has made a real and worthwhile difference (=6 points); "A great deal better, and a considerable improvement that has made all the diiference" (=7 points).
  The highest score corresponds to the most improvement in quality of life.
Evolution of quality of life (QoL): the Patient Benefit Index (PBI-L) | From baseline to 8 weeks of follow-up
  The evolution of QoL related to the lipedema is measured by the PBI-L self-questionnaire. It consists of 23 questions about different area: quality of life, physical, psychological. It consists of 2 questionnaires : before therapy and after therapy. The patient rates the extent to which the treatment objectives have been achieved. Questions are scaled from 0 'not important at all' to 4 'very important' with a response option 'does not apply to me'.
Evolution of lipedema-associated symptoms: Numeric Rating Scale (NRS) | From baseline to 8 weeks of follow-up
  The evolution of swelling, tightness, discomfort, heaviness, skin suppleness, fatigue due to lipedema is measured by NRS : 0 corresponds to no symptom and 10 to maximum symptom
Evolution of limb volume : tape perimeter measurements | From baseline to 8 weeks of follow-up
  The evolution of limb volume is measured by tape perimeter measurements taken from the dorsum of the foot and repeated for every 4 cm proximally until the root of the limb.
Evolution of skin tissue moisture : Moisture Meter | From baseline to 8 weeks of follow-up
  Changes in skin tissue moisture content are assessed by the Moisture Meter (Delfin Technologies Ltd, Finland).
Garment pressure : PicoPress | Baseline and 8 weeks of follow-up
  The pressure under the garment is measured by the Picopress. The PicoPress instrument is a portable digital gauge that measures the pressure exerted by a garment. The pressure detected by the transducer is displayed in Newton.
Evolution of inflammatory biological biomarker : C-reactive protein | From baseline to 8 weeks of follow-up
  The evolution of inflammatory biological biomarker : C-reactive protein (CRP) is measured from blood sample collection. The rate will be evaluated in milligrams per liter
Evolution of fat distribution: Waist to hip ratio | From baseline to 8 weeks of follow-up
  The evolution of fat distribution is calculated via the Waist-to-hip Ratio (WHR= waist circumference / hip circumference) and the Waist-to-Height-Ratio (WHtR= waist circumference / height).
Evolution of weight: BMI | From baseline to 8 weeks of follow-up
  The evolution of Body Mass Index (BMI) is calculated via the ratio Weight/(Size)2
Device safety | From baseline to 10 weeks
  The safety of the device is assessed by describing the adverse events (AEs) and serious adverse events (SAEs) that occur throughout the study.
Compliance to treatment | From baseline to 10 weeks
  The compliance to treatment (day and night) is reported by the physician according to the patient diary. The compliance is measured in average number of days that the device is worn.
Satisfaction about the device | 8 weeks, 10 weeks
  Patient's satisfaction with regards to the device is measured by a specific self-questionnaire given to the patient. The questionnaire is mainly focused on product positioning, comfort, stiffness with a 4 level-answer (example: very satisfied, satisfied, unsatisfied, very unsatisfied).

CONTACTS AND LOCATIONS:
Locations (1):
- La Fe University and Polytechnic Hospital, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alwardat N, Di Renzo L, Alwardat M, Romano L, De Santis GL, Gualtieri P, Carrano E, Nocerino P, De Lorenzo A. The effect of lipedema on health-related quality of life and psychological status: a narrative review of the literature. Eat Weight Disord. 2020 Aug;25(4):851-856. doi: 10.1007/s40519-019-00703-x. Epub 2019 May 6. PMID 31062201
- [Background] Esmer M, Schingale FJ, Unal D, Yazici MV, Guzel NA. Physiotherapy and rehabilitation applications in lipedema management: A literature review. Lymphology. 2020;53(2):88-95. PMID 33190432
- [Background] Forner-Cordero I, Forner-Cordero A, Szolnoky G. Update in the management of lipedema. Int Angiol. 2021 Aug;40(4):345-357. doi: 10.23736/S0392-9590.21.04604-6. Epub 2021 Apr 19. PMID 33870676
- See also: Related Info — https://lipedemaworldalliance.com/